CLINICAL TRIAL: NCT07234149
Title: Comparison of Color Stability, Bonding Time, and White Spot Lesion Between Flowable Nanocomposite and Packable Microhybrid Composite Used for Clear Aligner Attachments: A Split-Mouth Randomized Clinical Trial
Brief Title: Tooth Discoloration and Chairside Handling Time (Bonding-Debonding) in Flowable Versus Packable Composites for Clear Aligner Bonded Attachments: A Randomized Clinical Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sulaimani (Other)
Responsible Party: Principal Investigator, Elaf Hussein Hasan, MSc Student in Orthodontics, Ministry of Health, Iraq
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: USulaimani-Ortho-Aligner-2025; MSc-Ortho-Aligner-Study-2025; (Other: College of Dentistry, University of Sulaimani; Research Ethics Committee, College of Dentistry, University of Sulaimani)
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Clear Aligner Orthodontic Treatment; Composite Attachment; Color Stability of Enamel
Keywords: Composite Attachment Flowable Nanocomposite Packable Microhybrid Composite

STUDY DESIGN:
Intervention Model Description: Split-mouth randomized clinical trial in which each participant receives both interventions on opposite quadrants.
Who Masked: Outcomes Assessor
Masking Description: Single-blind design: the outcome assessor will be blinded to the type of composite used on each quadrant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- packable microcomposite (Group A) (Experimental): Participants will receive packable microcomposite attachments (e.g., GC G-ænial Universal ) on one side of the dental arc attachments on one quadrant of the dental arch for clear aligner therapy. Color change, bonding/debonding time, and enamel roughness will be assessed
  Interventions: Device: Packable Microhybrid Composite Resin
- flowable nanohybrid Composite (Group B) (Active Comparator): Participants will receive flowable nanocomposite (e.g., GC aligner connect ) attachments on the opposite quadrant of the same dental arch.Color change, bonding/debonding time, and enamel roughness will be assessed.
  Interventions: Device: flowable nanohybrid Composite Resin

INTERVENTIONS:
Device: flowable nanohybrid Composite Resin — A flowable nanocomposite (e.g., GC aligne connect) used to fabricate clear aligner attachments on enamel surfaces for comparison
  Other Names: packable microhybrid composite
  Arms: flowable nanohybrid Composite (Group B)
Device: Packable Microhybrid Composite Resin — Packable microhybrid composite resin used to fabricate clear aligner attachments.
  Arms: packable microcomposite (Group A)

SUMMARY:
This randomized split-mouth clinical trial aims to compare two different composite materials used for bonding attachments in clear aligner orthodontic therapy. Twenty adult participants with Class I malocclusion and mild crowding will receive flowable nanocomposite attachments on one side of the dental arch and packable microhybrid composite attachments on the opposite side. The primary outcome is the color change (ΔE) of the enamel surface after attachment removal, measured by a spectrophotometer (VITA Easyshade). Secondary outcomes include bonding and debonding time and changes in enamel surface roughness before and after treatment. The study will be conducted at the Orthodontic Department, College of Dentistry, University of Sulaimani. The goal is to determine which composite material provides better color stability, easier handling, and minimal impact on enamel surface characteristics during clear aligner therapy.

DETAILED DESCRIPTION:
Clear aligner therapy has become a popular alternative to conventional fixed orthodontic appliances due to its superior esthetics and comfort. However, the efficiency of aligner treatment often depends on the proper use of composite attachments that enhance tooth movement and retention. Different composite resins are used for this purpose, but their optical stability and effect on enamel integrity after removal remain concerns.

This prospective, split-mouth randomized clinical trial compares a flowable nanocomposite and a packable microhybrid composite used for clear aligner attachments. Each participant will receive both materials in opposite quadrants to minimize inter-individual variability. Outcomes will include enamel color change (ΔE CIE Lab* values), bonding/debonding time, and surface roughness assessment using digital and optical analysis methods.

The study hypothesis is that the flowable nanocomposite will exhibit superior color stability and faster handling time, with comparable enamel surface effects to the packable composite. Results from this trial may help establish standardized protocols for attachment material selection in clinical orthodontic practice.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18-40 years.
* patients with class l malocclusion with in which there treatment will be completed in 6 month .
* Completed clear aligner therapy and scheduled for attachment debonding at the study clinic.
* Permanent teeth with intact buccal enamel at assessment sites.
* No caries, restorations, cracks, fluorosis, or hypoplasia on assessed surfaces.
* No bleaching within 6 months prior to baseline.
* Good general health (ASA I-II) and able to provide written informed consent.
* Satisfactory oral hygiene and gingival health (e.g., GI ≤ 1).
* Willing and able to complete measurements: spectrophotometric shade (CIE L*, a*, b*), photographs/scans, and VAS for pain/discomfort.
* Available for all visits and follow-up assessment.

Exclusion Criteria:

* Patients younger than 18 or older than 40 years.
* Patients presenting with severe or very severe anterior crowding (LII > 6 mm) or spacing will exclude from the study. Cases with posterior crossbites, open bites, or skeletal discrepancies
* Presence of systemic diseases (ASA > II) that may affect healing, pain perception, or enamel quality.
* Teeth with caries, restorations, fractures, enamel cracks, fluorosis, hypoplasia, or discolorations on the buccal surfaces at assessment sites.
* Patients who have undergone tooth bleaching within the last 6 months.
* History of major dental surgery or trauma in the study region.
* Patients with poor oral hygiene or gingival inflammation (GI > 1).
* Pregnant or lactating women.
* Patients with allergy or hypersensitivity to composite resins or dental adhesives.
* Individuals unable to provide informed consent or not willing to comply with study visits.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-12-16 (Estimated)

PRIMARY OUTCOMES:
Change in Tooth Color (ΔE) After Attachment Removal | Baseline (before bonding) and after attachment removal
  The color change (ΔE) of the enamel surface will be measured using a VITA Easyshade spectrophotometer based on CIE Lab* values before bonding and after debonding of the attachments. A ΔE value ≥ 3.3 will be considered clinically perceptible.

CONTACTS AND LOCATIONS:
Overall Officials: Ali I Ibrahim, Principal Investigator — College of Dentistry, University of Sulaimani.
Locations (2):
- Iraq (2):
  - Private Orthodontic Clinic - Kirkuk, Kirkuk, Kirkuk Governorate
  - Private Orthodontic Clinic - Kirkuk, Kirkuk, Province

IPD SHARING:
Plan to Share IPD: No
ot applicable. Individual participant data will not be shared. Only summarized results will be published.

REFERENCES:
- [Result] Lin S, Huang L, Li J, Wen J, Mei L, Xu H, Zhang L, Li H. Assessment of preparation time and 1-year Invisalign aligner attachment survival using flowable and packable composites. Angle Orthod. 2021 Sep 1;91(5):583-589. doi: 10.2319/063020-598.1. PMID 33848325